CLINICAL TRIAL: NCT05393986
Title: An Open-Label, Single-Arm, Dose-Exploration Study to Evaluate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetics of CT048 in Subjects With Advanced Solid Tumors
Brief Title: Claudin18.2-redirected Chimeric Antigen Receptor T Cells With Co-expression of Cytokines in Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT048-CG4001
Record Dates: First submitted 2022-05-13; First posted 2022-05-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Gastric Adenocarcinoma; Pancreatic Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Claudin18.2; CAR-T cell therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: CAR-CLDN18.2 T-Cells (CT048) (Experimental): The subjects will be initially enrolled in the lymphodepletion cohort. Subsequent subjects will be enrolled in the non-lymphodepletion cohort after reviewing the data in the lymphodepletion cohort.
  Interventions: Drug: CT048 Autologous Injection (CT048)

INTERVENTIONS:
Drug: CT048 Autologous Injection (CT048) — up to 3 times CT048 Autologous Injection infusion
  Other Names: CT048 Autologous CAR T-cell Injection

SUMMARY:
An Open-Label, Single-Arm, Dose-Exploration Study to Evaluate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetics of CT048 in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is an open-label, single-arm, dose-escalation and dose-expansion, single/multiple infusion(s) exploratory study to evaluate the safety, tolerability, PK/PD and preliminary efficacy of CT048 in patients with advanced CLDN18.2+ solid tumors who had failed to at least 1 prior line of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, male or female;
2. Estimated life expectancy > 12 weeks;
3. Pathologically/histologically confirmed diagnosis of advanced G/GEJ adenocarcinoma or pancreatic cancer or other digestive system malignancies G/GEJA: refractory to or intolerable of at least 2 prior lines of treatment; HER2+ subjects must be refractory or intolerable of anti-HER2 treatment PC: refractory to or intolerable of at least 1 prior line of treatment;
4. Positive expression of CLDN18.2 in tumor tissue specimens;
5. According to the RECIST 1.1, there is measurable or unmeasurable tumor lesions;
6. ECOG physical status score 0 ~ 1 at screening, within 24 hours prior to apheresis;
7. Sufficient venous access for leukapheresis (central venous catheter)
8. Subjects should have adequate organ functions before screening :
9. Women of childbearing age (WOCB) be willing to use effective and reliable method of contraception (annual failure<1%) for at least 1 year after last infusion, and must refrain from donating sperms/eggs
10. Men who have actively sexual intercourse with women with child-bearing potential, must agree to use barrier-based contraception if they have no vasectomy. Moreover, all men are absolutely forbidden to donate sperm within 1 year after receiving the last infusion.

Exclusion Criteria:

1. High risks that may cause bleeding or perforation;
2. CNS metastasis, with or without related symptoms;
3. The presence of extensive lung metastases, or extensive liver metastases, or extensive bone metastases
4. History or current unstable or active digestive ulcers, gastrointestinal (GI) bleeding, GI obstruction;
5. Anti-tumor treatment for the investigational disease; treatment with anti-PD-1/PD-L1, anti-CTLA4, and any other immunotherapy or investigational therapy；
6. Prior treatment with any genetically modified cell therapy;
7. Treatment with systemic corticosteroids within 7 days prior to leukapheresis;
8. Prior solid organ transplantation, or allogeneic stem cell, or in the waiting list for organ transplantation;
9. Major surgical procedure or serious wound within 4 weeks prior to leukapheresis, or anticipation of need for a major surgical procedure during the study;
10. Positive serological tests of HIV, syphilis or HCV (subjects with positive HCV antibody but are negative for HCV RNA are eligible);
11. Any active or severe infection, incl. but not limited to active tuberculosis, HBV infection, etc.;
12. Active autoimmune disease;
13. Uncontrolled significant cardiovascular disease, pulmonary disease or CNS disease
14. History of malignancy other than investigational diseases within 3 years, with the exception of malignancies with a negligible risk of metastasis or death;
15. Pregnancy or lactating women;
16. History of allergic anaphylactic reactions to immunotherapy, and/or tocilizumab, cyclophosphamide, fludarabine or nab-paclitaxel, and/or CT048 components, or other history of severe allergic anaphylactic reactions ；
17. Blood oxygen saturation ≤95% before leukapheresis;
18. AEs from previous treatment that have not recovered to CTCAE ≤ grade 1, excluding hair loss, pigmentation, and other tolerable events and laboratory abnormalities permitted by the protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days of single infusion
  Safety
Maximum tolerated dose | 28 days of single infusion
  Tolerability

SECONDARY OUTCOMES:
Nature, incidence, severity and seriousness of TEAEs, TRAEs and AESI; graded according to the NCI-CTCAE (Version 5.0) or ASTCT | 1 year
  Adverse events occurring through 24 weeks and 12 months post CT048 indusion, such as abnormalities or changes in laboratory tests, physical examinations, vital signs, etc.
Pharmacokinetics(the number of CAR copies and CAR persistence duration in peripheral blood) | 1 year
  CAR-CLDN18.2 DNA in peripheral blood detected by q-PCR at each visit after each infusion
Antitumor efficacy-Overall response rate (ORR), Duration of response (DOR), Disease control rate (DCR) | 1 year
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the subjects should confirm it no less than 6 weeks after the first evaluation
Antitumor efficacy-Duration of response (DOR) | 1 year
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause
Antitumor efficacy-Disease control rate (DCR) | 1 year
  The number of cases in which response are achieved from the start of cell infusion/the total number of evaluable cases (%).
Antitumor efficacy-Progression-free survival | 1 year
  The period from the date of leukapheresis to the first recorded tumor progression or death of any cause, whichever occurs first (ITT).
Antitumor efficacy-Overall survival (OS) | 2 years
  The period from the date of leukapheresis to death of any cause (ITT). The period from the date of first CT048 infusion to death of any cause (mITT).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD,phD, Principal Investigator — Department of GI Oncology, Peking University Cancer Hospita
Locations (1):
- Beijing Cancer Hospital, Beijing, China, Beijing, China

IPD SHARING:
Plan to Share IPD: No